CLINICAL TRIAL: NCT04281069
Title: Diabetes Type 2 in the Eastern Region of Morocco , Towards an Evidence-based Multidisciplinary Lifestyle Approach in Diabetes Type 2
Brief Title: Diabetes Type 2 in the Eastern Region of Morocco
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Artesis Plantijn University College, Antwerp (Unknown); Université Mohammed Premier, Oujda (Unknown); Vliruos (Unknown)
Responsible Party: Principal Investigator, Van Rompaey Bart, associated professor, Universiteit Antwerpen
Other Study IDs: OZ7880VLIR-S
Record Dates: First submitted 2019-02-15; First posted 2020-02-24 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Quality of Life; Diabetes Mellitus, Type 2; Adherence, Medication; Diet Habit
Keywords: diabetes mellitus type 2; quality of life; interdisciplinary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients visiting the "centre de santé": Women visiting to the selected health centres in the Oujda province will be invited to participate

SUMMARY:
This South Initiative is the first step towards a long-term general objective that aims to improve the manage-ment of type 2 diabetes (T2D) and concurrently create jobs for health professionals in Eastern Morocco by developing a multidisciplinary approach in the management of T2D, based upon international guidelines but adapted to the regional socio-economic and cultural context, and with a focus on empowerment of Muslim women.

The intermediate results of this SI project proposal are: 1) Facilitators and perceived barriers in female patients with T2D towards change to a healthier lifestyle are known. 2) Characteristics of patients with T2D in the region of Oujda (prevalence, lifestyle, age, gender,…) are analysed. 3) Master and bachelor students have gained experience by participating to relevant research. 4) All involved stakeholders shared existing and newly ac-quired knowledge and expertise. 5) Facilitators and perceived barriers in health professionals of different disciplines to work together in the management of T2D are known.

DETAILED DESCRIPTION:
The ultimate objective is to help improve the quality of life and well-being of people living with diabetes in the Oujda region.

This 2-year project will tackle the prerequisites and optimise the conditions needed to start a larger (TEAM) project. Afterwards, in the larger long-term (TEAM) project we will study the cost-of illness of T2D in Oujda, the effect of a cultural-sensitive multidisciplinary intervention for T2D and the cost-effectiveness of such an intervention. In doing so we hope to provide not only arguments from a health perspective for such an approach, but also from a quality of life and economic point of view. This is needed to persuade political decision makers to invest in sustainable innovation in health care. This could open the job market for many young physiotherapists, nutritionists and occupational therapists in health centres and primary care.

The specific objectives of this 2-year SI project are 1) to know the characteristics of T2D patients in Oujda and their perceived barriers and benefits towards participation in a lifestyle program and 2) to improve communication and cooperation between health professionals of different disciplines treating patients with T2D.

The intermediate results of this 2-year project are well defined and feasible (Annex 4). The two years of the SI project will be devoted to gathering information from diabetic women as well as from health profes-sionals, to creating a platform and to strengthening research capacities. The changes needed to reach the SI project outputs are related to 1) knowledge/capacity and 2) attitude/behaviour.

ELIGIBILITY:
Inclusion Criteria:

* women
* visiting the 35 local health centres and the CRD in Oujda
* adult
* Moroccan

Exclusion Criteria:

* male
* no informed consent

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: step 1) all women, diagnosed with diabetes or not step 2) adults diagnosed with diabetes type 2
Sampling Method: Non-Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
glycaemia | first year
  the concentration of glucose in the blood

SECONDARY OUTCOMES:
Hemoglobin A1c | first year
  The concentration of hemoglobin A1c in the blood shows the average level of blood sugar over the past 2 to 3 months.

OTHER OUTCOMES:
systolic and diastolic blood pressure | first year
  common systolic and diastolic assessment of blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Université Mohammed Premier Oujda (UMP) Faculté des Sciences, Département de Biologie, Oujda, Oujda Angad, Morocco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollard TM, Guell C. Assessing physical activity in Muslim women of South Asian origin. J Phys Act Health. 2012 Sep;9(7):970-6. doi: 10.1123/jpah.9.7.970. PMID 22971888
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Abuyassin B, Laher I. Diabetes epidemic sweeping the Arab world. World J Diabetes. 2016 Apr 25;7(8):165-74. doi: 10.4239/wjd.v7.i8.165. PMID 27114755
- [Background] Palmer AJ, Roze S, Valentine WJ, Spinas GA, Shaw JE, Zimmet PZ. Intensive lifestyle changes or metformin in patients with impaired glucose tolerance: modeling the long-term health economic implications of the diabetes prevention program in Australia, France, Germany, Switzerland, and the United Kingdom. Clin Ther. 2004 Feb;26(2):304-21. doi: 10.1016/s0149-2918(04)90029-x. PMID 15038953
- [Background] Lindstrom J, Peltonen M, Eriksson JG, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS). Improved lifestyle and decreased diabetes risk over 13 years: long-term follow-up of the randomised Finnish Diabetes Prevention Study (DPS). Diabetologia. 2013 Feb;56(2):284-93. doi: 10.1007/s00125-012-2752-5. Epub 2012 Oct 24. PMID 23093136